CLINICAL TRIAL: NCT00241384
Title: Low Dose Supplemental External Radiation With PD-103 Versus PD-103 Alone For Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Schiffler Cancer Center (Other)
Collaborators: Theragenics (Unknown); University of Washington (Other)
Responsible Party: Principal Investigator, Gregory Merrick, M.D., Medical Director, Schiffler Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-8-10
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
Keywords: Prostatic Cancer; Brachytherapy; Prostatic neoplasm; Radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Palladium-103

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pd-103 with 20Gy External Beam (Active Comparator): Pd-103 with 20Gy External Beam
  Interventions: Procedure: External beam radiation
- Pd-103 alone (Active Comparator): Pd-103 alone
  Interventions: Procedure: Pd-103

INTERVENTIONS:
Procedure: External beam radiation
  Arms: Pd-103 with 20Gy External Beam
Procedure: Pd-103
  Arms: Pd-103 alone

SUMMARY:
The primary purpose of this study is to evaluate two treatment regimens for prostate cancer, prostate implant with 20 Gy of external beam radiation therapy versus prostate implant with 0 Gy of external beam radiation therapy. Patients diagnosed with intermediate risk prostate cancer between the ages of 40 and 80 who have chosen brachytherapy with or without external beam radiation therapy as their intended treatment will be eligible and will be offered participation.

DETAILED DESCRIPTION:
Approximately 250,000 men are currently diagnosed with prostatic cancer in the United States each year. Of those, 70% have stage T1 or T2 disease (apparently limited to the prostate gland). Clinically localized prostate cancer is a spectrum of disease, ranging from good prognosis to poor prognosis. Patients with a PSA above 10 ng/ml or Gleason score of 7 to 10 are referred to as intermediate risk, with approximately an 80% chance of cure.

Implantation of radioactive sources directly into the prostate (brachytherapy) delivers a high, localized radiation dose while sparing most the of the bladder and rectum. Brachytherapy is well established for other tumor sites, and has become a standard treatment for prostate cancer.

Establishing that a good quality implant alone is as effective as implant plus beam radiation will allow us to routinely drop the use of beam radiation, a change in policy that will decrease the risk of some complications, will be more convenient for patients, and will lower treatment costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated prostatic cancer.
* Must have PSA 10-20 ng/ml, Gleason 7 to 9

Exclusion Criteria:

* Patients with proven regional lymph node involvement will be excluded.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2005-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Serial PSA : 6, 12, 18 and 24 months and then yearly. | 6, 12, 18 and 24 months and then yearly
  Serial PSA : 6, 12, 18 and 24 months and then yearly.
Post treatment biopsies in those with persistently elevated | as needed
  Post treatment biopsies in those with persistently elevated
PSA which is suggestive of residual tumor. | as needed
  PSA which is suggestive of residual tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory S Merrick, MD, Principal Investigator — Schiffler Cancer Center, Wheeling, WV; Kent E Wallner, MD, Study Chair — University of Washington VA Center
Locations (2):
- United States (2):
  - Veterans Administration Puget Sound Health Care System, Seattle, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia

REFERENCES:
- [Background] Bartolini R, Dattoli G, Giannessi L, Mezi L, Renieri A, Migliorati M, Bruni C, Couprie ME, Garzella D, Orlandi G. Saturation and electron-beam lifetime in a storage ring free-electron laser. Phys Rev E Stat Nonlin Soft Matter Phys. 2004 Mar;69(3 Pt 2):036501. doi: 10.1103/PhysRevE.69.036501. Epub 2004 Mar 4. PMID 15089421
- [Background] Blasko JC, Grimm PD, Sylvester JE, Badiozamani KR, Hoak D, Cavanagh W. Palladium-103 brachytherapy for prostate carcinoma. Int J Radiat Oncol Biol Phys. 2000 Mar 1;46(4):839-50. doi: 10.1016/s0360-3016(99)00499-x. PMID 10705004
- [Background] Critz FA, Williams WH, Levinson AK, Benton JB, Holladay CT, Schnell FJ Jr. Simultaneous irradiation for prostate cancer: intermediate results with modern techniques. J Urol. 2000 Sep;164(3 Pt 1):738-41; discussion 741-3. doi: 10.1097/00005392-200009010-00028. PMID 10953137
- [Background] Merrick GS, Butler WM, Galbreath RW, Lief JH. Five-year biochemical outcome following permanent interstitial brachytherapy for clinical T1-T3 prostate cancer. Int J Radiat Oncol Biol Phys. 2001 Sep 1;51(1):41-8. doi: 10.1016/s0360-3016(01)01594-2. PMID 11516849
- [Background] Blue E. Letting go of Ben. Nurs Spectr (Wash D C). 1999 Mar 8;9(5):20. No abstract available. PMID 10562177
- [Background] Potters L, Cao Y, Calugaru E, Torre T, Fearn P, Wang XH. A comprehensive review of CT-based dosimetry parameters and biochemical control in patients treated with permanent prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2001 Jul 1;50(3):605-14. doi: 10.1016/s0360-3016(01)01473-0. PMID 11395226
- [Background] Blasko JC, Ragde H, Schumacher D. Transperineal percutaneous iodine-125 implantatio for prostatic carcinoma using transrectal ultrasound and template guidance. Endo/Hypertherm 1987;3:131-39.
- [Background] Wallner K, Merrick G, Butler W, Sheretz T, Sutlief S, Cavanagh W, et al. 20 Gy versus 44 Gy supplemental beam radiation combined with Pd-103 prostate brachytherapy: early results from a prospective randomized multicenter trial (submitted)2004.
- [Background] Prestidge BR, Hoak DC, Grimm PD, Ragde H, Cavanagh W, Blasko JC. Posttreatment biopsy results following interstitial brachytherapy in early-stage prostate cancer. Int J Radiat Oncol Biol Phys. 1997 Jan 1;37(1):31-9. doi: 10.1016/s0360-3016(96)00390-2. PMID 9054874
- [Background] Zietman AL, Tibbs MK, Dallow KC, Smith CT, Althausen AF, Zlotecki RA, Shipley WU. Use of PSA nadir to predict subsequent biochemical outcome following external beam radiation therapy for T1-2 adenocarcinoma of the prostate. Radiother Oncol. 1996 Aug;40(2):159-62. doi: 10.1016/0167-8140(96)01770-7. PMID 8884970